CLINICAL TRIAL: NCT04378998
Title: Is Acupuncture Able to Reduce Nausea and Vomiting in the Terminal Ill Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-291-14
Record Dates: First submitted 2020-04-28; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Terminal Illness
Keywords: Acupuncture; Nausea; Vomiting; Palliative care
MeSH Terms: conditions — Nausea; Vomiting | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): The intervention group received usual care plus acupuncture for three days. The acupuncture spots: Pericardium-6, Stomach-36, Liver-3 and Ying Tang were used.
  Interventions: Other: Acupuncture
- Usual care (No Intervention)

INTERVENTIONS:
Other: Acupuncture — The intervention group received usual care plus acupuncture for three days. The acupuncture spots: Pericardium-6, Stomach-36, Liver-3 and Yin Tang were used. The control group received usual care.
  Arms: Acupuncture

SUMMARY:
A comparative effectiveness research design was used. The sample size was calculated to 136 patients, who were randomized to an intervention group and a control group respectively. The patients were terminal ill patients enrolled to three in-bed hospices in Denmark and nausea and vomiting were measured using EORTC QlQ-c15-PAL (European Organisation for Research and Treatment of Cancer, Quality of Life Questionaire, core 15, Palliation)

DETAILED DESCRIPTION:
The terminal ill patient is suffering from many different symptoms. In total 70% are suffering from nausea and vomiting due to the wide spread of cancer or due to side effects of treatment. Often the antiemetic's are not able to reduce symptoms to a level that enable the patient to experience quality in life in the last days of his life. The investigators had some experience with acupuncture as a complementary therapy but the investigators wanted more systematically to investigate if acupuncture is able to reduce the terminal ill patient´s nausea and vomiting. Literature show that acupuncture is able to reduce nausea and vomiting in patients receiving chemotherapy, but there is no literature that support the ability of acupuncture to reduce nausea and vomiting in the terminal ill patient.

The purpose of this study was to generate evidence based knowledge close to practice regarding the effect of acupuncture in reducing nausea and vomiting in the terminal ill patient.

Participants:

Terminal ill patients suffering from nausea and/or vomiting

Interventions:

The intervention group received usual care plus acupuncture for three days. The acupuncture spots: Pericardium-6, Stomach-36, Liver-3 and Yin Tang were used. The control group received usual care.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate due to cognitive ability
* Nausea
* Admitted to in-bed hospice

Exclusion Criteria:

* Not able to participate due to cognitive impairment
* Lymphedema in the area of acupuncture site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-01-25 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Change in nausea score | Change in nausea score from before intervention to three day after the intervention
  Using EORTC QLQ-c15-PAL, the nausea item. Values: not at all, a little, quite a bit, very much. Very much is the worse outcome
Change in vomiting | Change in vomiting from before intervention to four day after the intervention
  Unit of measure: Incidence of vomiting using the outcome measure question: Yes or No

IPD SHARING:
Plan to Share IPD: No